CLINICAL TRIAL: NCT03544710
Title: The Impact of Preoperative Bathing With Chloroxylenol on the Incidence of Post Caesarean Section Surgical Site Infection at Mbarara Regional Referral Hospital: A Randomized Controlled Trial
Brief Title: Impact of Preoperative Bathing on Post Caesarean Section Surgical Site Infection
Acronym: SSI-MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08/08-17
Record Dates: First submitted 2018-05-20; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Cesarean Wound Disruption With Postnatal Complication
Keywords: surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Anti-Infective Agents, Local

STUDY DESIGN:
Intervention Model Description: The participants in the bathing arm were each given warm water and a tablet of soap containing chloroxylenol antiseptic and they were asked to bathe using it within at most two hours prior to the surgery. After bathing, the participants were given a clean theatre gown to put on, after which they were taken through the routine pre-operative preparation procedures according to the existing ward protocol.
  The participants in the control arm were only taken through the routine preoperative preparation procedures according to the existing ward protocol
Who Masked: Outcomes Assessor
Masking Description: Mothers scheduled to deliver by emergency Caesarean section were randomly assigned to either bathing or routine care arms in a ratio of 1:1. We did simple randomization to either bathing or routine care arm without any blocks. We generated patient group assignments using the computer algorithm (computer-generated list of random numbers). The research assistant who enrolled mothers into the study assigned the study arm by checking from the list of random numbers. The research assistant and the PI, who were on the outcomes assessment arm was not allowed to ask the study participant concerning the allocation arm. Single blinding of PI and one of the research assistants assessing outcomes was done to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing (Experimental): Intervention was Preoperative bathing with antiseptic. Given warm water and a tablet soap containing chloroxylenol antiseptic. Asked to bathe under supervision for standardization. Given a clean theatre gown to put on. Taken through the routine pre-operative preparation procedures which involved; Putting an intravenous cannula; administering prophylactic antibiotics. Administering intravenous normal saline 1 liter. taking off a blood sample (3mls) for blood grouping and cross matching. Putting urethral catheter for drainage of urine, Getting an informed consent from the client for the procedure to be done. Informing the theatre team.
  Interventions: Other: preoperative bathing with antiseptic
- No bathing (No Intervention): No intervention done for participants in this arm. They go through the routine ward procedure as below.
  Putting an intravenous cannula; administering prophylactic antibiotics. Administering intravenous normal saline 1 liter. taking off a blood sample (3mls) for blood grouping and cross matching. Putting urethral catheter for drainage of urine, Getting an informed consent from the client for the procedure to be done. Informing the theatre team.

INTERVENTIONS:
Other: preoperative bathing with antiseptic — Preoperative bathing with antiseptic was done as follows; Given warm water and a tablet soap containing chloroxylenol antiseptic.
  Asked to bathe under supervision for standardization. Given a clean theatre gown to put on. Taken through the routine pre-operative preparation procedures which involved; Putting an intravenous cannula; administering prophylactic antibiotics. Administering intravenous normal saline 1 liter. taking off a blood sample (3mls) for blood grouping and cross matching. Putting urethral catheter for drainage of urine, Getting an informed consent from the client for the procedure to be done. Informing the theatre team.
  Arms: Bathing

SUMMARY:
Surgical site infection (SSI) is the commonest hospital-acquired infection globally, and prevalence is much higher in the low-income countries. Caesarean delivery carries a 5-20 fold risk for developing postpartum sepsis. SSIs cause significant morbidity, prolonged hospitalization and mortality. Simple and inexpensive interventions like preoperative bathing need to be studied, to assess their impact on surgical site infection rates.

DETAILED DESCRIPTION:
Caesarean delivery is the single-most important risk factor for postpartum pregnancy associated infections carrying a 5 to 20-fold increase in the risk of developing sepsis. Research done in MRRH showed a post-surgery wound sepsis prevalence of 82% on all surgical wards in the hospital and the prevalence of post caesarean section wound infection at MRRH is 15.5%. At MRRH, surgical site infections remain a substantial cause of morbidity, prolonged hospitalization and mortality. SSI is associated with a mortality rate of 3%, and 75% of SSI associated deaths are directly attributable to the SSIs. Universal practices like preoperative bathing of patients are currently not being practiced at MRRH and thus their impact on reducing the burden can only be speculated upon. The aim of this study was to assess the impact of preoperative bathing with chloroxylenol antiseptic on the incidence of post caesarean section surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* All mother scheduled for delivery by emergency C/S at MRRH during the study period.

Exclusion Criteria:

* Women who declined to consent.
* Women with obvious evidence of infection, like fever, foul-smelling liquor, or those already on antibiotics for reasons other than preoperative prophylaxis.
* Women in whom delivery was indicated to occur within less than 30 minutes, like in fetal distress, obstructed labor, pulsatile cord prolapse, or ruptured uterus.
* Women who could not communicate and give information for the study and those who do not have a working telephone contact.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Clinical diagnosis was made based on the CDC- 2013 definition of SSI

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lukabwe, MD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after obtaining all necessary permission

REFERENCES:
- [Derived] Lukabwe H, Kajabwangu R, Mugisha D, Mayengo H, Munyanderu B, Baluku A, Manyang A, Lapat JJ, Banya F, Kayondo M, Mayanja R, Muhumuza J, Bajunirwe F, Ngonzi J. Effectiveness of preoperative bath using chloroxylenol antiseptic soap on the incidence of post emergency cesarean section surgical site infection at Mbarara Regional Referral hospital, Uganda: a randomized controlled trial. Pan Afr Med J. 2022 Feb 2;41:92. doi: 10.11604/pamj.2022.41.92.23687. eCollection 2022. PMID 35465375
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252